CLINICAL TRIAL: NCT06248047
Title: Vessel-sparing Technique Versus Conventional Repair of Pelvic Fracture Urethral Injury: A Prospective Comparative Study
Brief Title: Vessel-sparing Technique Versus Conventional Repair of PFUI: A Prospective Comparative Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Hosam Mahdy, teaching assistant of urology, Assiut University
Other Study IDs: new urethroplasty technique
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Urethral Stricture, Male, Overlapping Sites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conventional repair: the patients will undergo repair with no regard to the vessels .then follow up by uroflow ,ascending urethrogram and penile doppler .
  Interventions: Procedure: uretheroplasty
- the new technique: the patients will undergo repair with sparing of the vessels .then follow up by uroflow ,ascending urethrogram and penile doppler .
  Interventions: Procedure: uretheroplasty

INTERVENTIONS:
Procedure: uretheroplasty — 4. When the bulb and bulbar urethra are exposed and before further dissection, the bulbar arteries are located using a directional doppler ultrasound stethoscope and a decision is made to sacrifice the artery with the lowest doppler signal to preserve the contralateral best artery. The bulbar urethra is then mobilized, circumferentially dissected and separated distally from the corpus cavernosum up to the penoscrotal angle to gain sufficient length for a tension-free end-to-end anastomosis without detachment of the bulb from the perineal body. If the dissection is not sufficient to bridge the gap,inter-corporal septal separation or even an inferior pubectomy are performed. The scarred tissue is removed completely, the proximal urethral segment is exposed as usual with spatulation of the healthy urethral ends and end-to-end anastomosis of the urethra over a silicon catheter is performed. No dissection is performed contralaterally at the bulb to preserve the artery of that side.

SUMMARY:
Pelvic fracture is associated with urethral injury in about 10% of patients . The common site of injury is at the bulbomembranous Junction and anastomotic urethroplasty with a tension free anastomosis remains the gold standard management for pelvic fracture urethral injury (PFUI) .

Traditional reconstruction of PFUI requires mobilization of the bulbar urethra to reach the prostatic apex with deep dissection of the spongiosum and detachment of the bulb from the perineal membrane at the site of the bulbomembranous urethral injury, a maneuver that requires division of the bulbar arteries . Then, the distal bulb and bulbar urethra will depend on retrograde blood flow through the glans and some perforating branches of the dorsal penile artery and this is usually sufficient to maintain good vitality of the spongiosum and urethra under normal circumstances .

When the distal blood supply to the urethra is compromised, either by congenital anomalies such a hypospadias, by previous surgery, or by the pre-existing pelvic fracture, the retrograde flow to the spongiosum is insufficient . In such cases, traditional anastomotic urethroplasty may result in ischemic bulbar necrosis, leading to a reconstructive failure and these patients usually fail to void soon after removal of the catheter, with subsequent retrograde urethrogram (RUG) showing a long bulbar urethral defect .

In 2007, Jordan et al described a modification to excision and primary anastomosis (EPA) in the proximal bulbar urethral strictures particularly post radical prostatectomy, which includes mobilizing and preserving the bulbar arteries with the continuity of the corpus spongiosum is maintained .

Gomez et al believed that vessel-sparing anastomotic urethroplasty is highly relevant in the PFUI scenario as it can theoretically help to avoid ischemic failure and cold glans syndrome improving sexual arousal. Consequently, they modified the standard reconstructive technique for PFUI by preserving bulbar arterial inflow .

So that, we decide to compare between vessel-sparing technique and conventional repair in management of PFUI through a prospective study.

ELIGIBILITY:
Inclusion Criteria:

- Adult male patients ≥ 18 years old with PFUI

Exclusion Criteria:

* Recurrent cases. • History of concomitant bladder neck injury

Ages: 18 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: patient with pelvis fracture type A , B and C , cystocathater .
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
UROFLOWMETERY | three months after the operation
  the speed and feasibility of micturition measured by non invasive pressure flow study Q max more than 10ml/sec
postmicturition residue | three months after the operation
  abdominal ultrasound done to evaluate PMR
Retrograde Urethrogram RUG | three months after the operation
  contrast study to evaluate and delineate the urethera

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Durrant JJ, Ramasamy A, Salmon MS, Watkin N, Sargeant I. Pelvic fracture-related urethral and bladder injury. J R Army Med Corps. 2013 Mar;159 Suppl 1:i32-9. doi: 10.1136/jramc-2013-000025. PMID 23631324
- [Background] Webster GD, Ramon J. Repair of pelvic fracture posterior urethral defects using an elaborated perineal approach: experience with 74 cases. J Urol. 1991 Apr;145(4):744-8. doi: 10.1016/s0022-5347(17)38442-2. PMID 2005693
- [Background] Kulkarni SB, Surana S, Desai DJ, Orabi H, Iyer S, Kulkarni J, Dumawat A, Joshi PM. Management of complex and redo cases of pelvic fracture urethral injuries. Asian J Urol. 2018 Apr;5(2):107-117. doi: 10.1016/j.ajur.2018.02.005. Epub 2018 Mar 2. PMID 29736373
- [Background] Gomez RG, Campos RA, Velarde LG. Reconstruction of Pelvic Fracture Urethral Injuries With Sparing of the Bulbar Arteries. Urology. 2016 Feb;88:207-12. doi: 10.1016/j.urology.2015.09.032. Epub 2015 Nov 23. PMID 26616094
- [Background] Gur U, Jordan GH. Vessel-sparing excision and primary anastomosis (for proximal bulbar urethral strictures). BJU Int. 2008 May;101(9):1183-95. doi: 10.1111/j.1464-410X.2008.07619.x. No abstract available. PMID 18399836